CLINICAL TRIAL: NCT04324801
Title: Aftereffects and Reliability of Two Homeostatic Plasticity Induction Protocols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Priscilla G. Wittkopf, Principal Investigator, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20190069
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): This is a within-subject repeated-measures design.
  Interventions: Other: Homeostatic plasticity induction using transcranial direct current stimulation

INTERVENTIONS:
Other: Homeostatic plasticity induction using transcranial direct current stimulation — Homeostatic plasticity will be induced in the left primary motor cortex using tDCS applied for 7 minutes followed by an interval of 3 minutes and another block of 5 minutes of stimulation

SUMMARY:
People suffering from chronic pain exhibit changes in the way the central nervous system processes pain. Some of the changes in the central nervous system are associated with how the brain adapts to the process of different stimuli. There are several physiological mechanisms that regulates how the brain adapts to changes and one of these mechanisms is called homeostatic plasticity (or equilibrium plasticity ). In healthy participants homeostatic plasticity mechanisms have been tested and considered normal, whereas in patients with chronic conditions, such as low back pain, this mechanism was shown to be dysfunctional. However, it is unknown when this difference in the pain system develops. It is possible that homeostatic mechanism becomes impaired over a period of time. Current studies have investigate a cohort of patients and there is a lack of longitudinal designs. In order to investigate the long-term effects of pain on homeostatic plasticity mechanisms it is important to first investigate the reliability of the methods. This study will investigate the reliability of two protocols of homeostatic plasticity induction.

DETAILED DESCRIPTION:
The aim of this study is to investigate the corticomotor excitability changes provoked by two homeostatic plasticity induction protocols, specifically the duration and the test-retest reliability of such corticomotor excitability changes.

A within-subject repeated-measures design will be used to evaluate the aftereffects and the reliability of two homeostatic plasticity induction protocols using cathodal transcranial direct current stimulation (tDCS) (experiment 1) and anodal tDCS (experiment 2). Each participant will take part in two experimental sessions during which homeostatic plasticity and corticomotor excitability will be induced and measured in the left primary motor cortex.

A sample size calculation was conducted using α of 0.05, β of 0.80 and effect size of 0.48 based on motor evoked potential (MEP) analysis of previous studies (Thapa, Schabrun, 2018, Thapa et al., 2018) resulting in a target of 13 participants. To account for differences in study designs and for the possibility of participant withdrawal/dropout, the investigators set target recruitment at 15 participants for each experiment.

Each participant will attend two identical experimental sessions on the same time in two consecutive days. During the experiment, participants will be seated comfortably with hands and arms at rest. First, the electromyography electrodes will be placed at the right hand muscle to be used for assessing the corticomotor excitability by recordings of motor evoked potentials by transcranial magnetic stimulation (TMS) on the left primary motor cortex. Then, the neoprene cap for tDCS on the left primary motor cortex will be mounted. The optimal scalp position (hot spot) for TMS stimulation will be identified and marked with a pen on the cap for standardisation. The corticomotor excitability in response to the homeostatic plasticity protocol (cathodal tDCS in experiment 1 or anodal tDCS in experiment 2) will be measured before and immediately post paradigm (time point 0-min), and then every 10 minutes for 70 minutes.

Homeostatic plasticity will be induced in the left primary motor cortex using tDCS applied for 7 minutes followed by an interval of 3 minutes and another block of 5 minutes of stimulation (Thapa, Schabrun, 2018, Thapa et al., 2018). A constant current of 1mA will be transmitted through the tDCS system (Starstim, Neuroelectrics, Barcelona, Spain), using two 3.14 cm2 Ag/AgCl gelled electrodes placed into holes of a neoprene cap corresponding to the international 10/10 EEG system, placed on participants head with the central Cz position aligned to the vertex of the head. In experiment 1 the cathode will be placed at C3 and return electrode placed at Fp2. In experiment 2 the anode will be placed at C3 and return electrode placed at Fp2.

Data distribution will be assessed using the Shapiro-Wilk test. A repeated measures analysis of variance (ANOVA) will be conducted on mean MEPs with factors Session (Day1 and Day2) and Time (baseline, 0 min, 10 min, 20 min, 30 min, 40 min, 50 min, 60 min, 70 min). A Greenhouse-Geisser correction will be used if Mauchly's test shows that sphericity cannot be assumed. Adjustments will be made for multiple post-hoc comparisons using the Bonferroni correction. Results will be interpreted according to the level of statistical significance p≤0.05 and effect size reported as partial eta squared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, aged between 18-60 years, right-handed and can speak and understand English.

Exclusion Criteria:

* Lack of ability to cooperate
* History or present chronic pain or current acute pain
* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Present and previous neurological disorders such as epilepsy, Alzheimer's disease, dementia, stroke, migraine and other headache disorders, multiple sclerosis, Parkinson's disease, neuroinfections, brain tumors and head trauma.
* Present or previous musculoskeletal disorders such as tendonitis, degenerative disc disease, mechanical back syndrome, and ruptured/herniated disc.
* Present or previous mental illnesses such as depression, bipolar disorder, and schizophrenia.
* Current use of medications that may affect the trial (e.g. analgesics, anti-inflammatories, anti-depressives)
* Contraindications to TMS application (history of epilepsy, metal implants in head or jaw, etc.)
* Failure to pass the tDCS screening questionnaire
* Failure to pass the "TASS questionnaire"

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Motor evoked potentials change from baseline | 0 minutes post homeostatic plasticity induction
Motor evoked potentials change from baseline | 10 minutes post homeostatic plasticity induction
Motor evoked potentials change from baseline | 20 minutes post homeostatic plasticity induction
Motor evoked potentials change from baseline | 30 minutes post homeostatic plasticity induction
Motor evoked potentials change from baseline | 40 minutes post homeostatic plasticity induction
Motor evoked potentials change from baseline | 50 minutes post homeostatic plasticity induction
Motor evoked potentials change from baseline | 60 minutes post homeostatic plasticity induction
Motor evoked potentials change from baseline | 70 minutes post homeostatic plasticity induction

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thapa T, Graven-Nielsen T, Chipchase LS, Schabrun SM. Disruption of cortical synaptic homeostasis in individuals with chronic low back pain. Clin Neurophysiol. 2018 May;129(5):1090-1096. doi: 10.1016/j.clinph.2018.01.060. Epub 2018 Feb 9. PMID 29472134
- [Background] Thapa T, Schabrun SM. Test-Retest Reliability of Homeostatic Plasticity in the Human Primary Motor Cortex. Neural Plast. 2018 Jun 10;2018:6207508. doi: 10.1155/2018/6207508. eCollection 2018. PMID 29983706
- [Background] Karabanov A, Ziemann U, Hamada M, George MS, Quartarone A, Classen J, Massimini M, Rothwell J, Siebner HR. Consensus Paper: Probing Homeostatic Plasticity of Human Cortex With Non-invasive Transcranial Brain Stimulation. Brain Stimul. 2015 May-Jun;8(3):442-54. doi: 10.1016/j.brs.2015.01.404. Epub 2015 Apr 1. PMID 26050599
- [Background] Fricke K, Seeber AA, Thirugnanasambandam N, Paulus W, Nitsche MA, Rothwell JC. Time course of the induction of homeostatic plasticity generated by repeated transcranial direct current stimulation of the human motor cortex. J Neurophysiol. 2011 Mar;105(3):1141-9. doi: 10.1152/jn.00608.2009. Epub 2010 Dec 22. PMID 21177994
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650